CLINICAL TRIAL: NCT03893032
Title: Enhancing Operational Performance in Healthy Rested Soldiers With Pharmacological Stimulants
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: United States Army Aeromedical Research Laboratory (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amanda Kelley, Research Psychologist, United States Army Aeromedical Research Laboratory
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: USAARL 2018-007; IRB M-10746
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Cognition
MeSH Terms: interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Modafinil 200mg (Experimental): single, 200 mg dose of modafinil
  Interventions: Drug: Modafinil 200mg
- mixed amphetamine salts (Experimental): single 10 mg dose of mixed amphetamine salts
  Interventions: Drug: mixed amphetamine salts
- placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Modafinil 200mg — single 200 mg dose
  Arms: Modafinil 200mg
Drug: mixed amphetamine salts — single 10 mg dose
  Arms: mixed amphetamine salts
Drug: Placebo — single oral-administration placebo tablet
  Arms: placebo

SUMMARY:
Considerable research has documented the optimization utility of stimulants in sleep deprived Soldiers and aviators, however, the research for enhancement purposes has demonstrated mixed results. One significant factor that may influence enhancement properties is general intelligence such that low performers exhibit stronger enhancement effects than high performers. The objective of this study is to determine whether stimulants (specifically, modafinil and Adderall) can enhance Soldier cognitive abilities and performance on military tasks. To do so, a within-subjects design will be employed using healthy, rested Soldiers and measuring performance on a set of basic cognitive assessments and operationally relevant tasks.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years old.
* Must have normal hearing, vision or corrected to normal vision, and cognitive function as determined by self-report
* Must have obtained at minimum 6 hours of sleep prior to all testing sessions, as assessed by actigraphy data and self-report. Should the actiwatch malfunction, reliance on self-report will suffice. If the subject does not meet this requirement, he will be asked to reschedule
* Must have refrained from consumption of stimulants (including caffeine) and over the counter medications which may induce drowsiness for a minimum of 16 hours prior to each test session, and nicotine, 8 hours, prior to all testing sessions, assessed by self-report.

Exclusion Criteria:

* Currently taking medications which induce drowsiness, such as over-the-counter antihistamines. Any self-medication will be assessed through self-report.
* No current medical conditions or medications affecting cognitive function or attention as determined by screening by study physician or medical practitioner
* Current or recent use (as determined by study physician or medical practitioner) of medications that may interact with the test articles. Determined by self-report and exclusion at the discretion of the study physician or medical practitioner.
* Any history of any attention deficit condition requiring medication. A history of any attention deficit condition with medication is disqualifying as the potential interactions with testing are unknown and would therefore produce a potential source of confounding or bias into the results of the study.
* Any history of psychological/psychiatric disorder.
* Any history of addiction or substance abuse as assessed through self-report.
* Any history of metabolic disorder such as dysthyriodism.
* Any history of significant cardiovascular disease or hypertension.
* Any history of hepatic or renal disorder.
* Females will be excluded given that the drugs administered could potentially negatively impact the very early stages of pregnancy.
* Any ingestion of substances that may interact with the test articles or potentially skew the results within the last 16 hours prior to testing including over-the-counter medications, supplements, etc. (see attached list to be reviewed with subject).

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-07-17 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
change from baseline in working memory performance | 2-hours post-dosing
  Digit span task
change from baseline in selective attention performance | 2-hours post-dosing
  Stroop test
change from baseline in sustained attention performance | 2-hours post-dosing
  Rapid Visual Information Processing Task
change from baseline in executive function performance | 2-hours post-dosing
  Digit symbol substitution task
change from baseline in marksmanship performance | 2-hours post-dosing
  number of targets acquired on marksmanship trainer

SECONDARY OUTCOMES:
change from baseline in impulsivity | 2-hours post-dosing
  Stop signal task - response inhibition
change from baseline in impulsivity | 2-hours post-dosing
  Continuous Performance test - rapid response initiation
change from baseline in risk-taking behavior | 2-hours post-dosing
  Evaluation of Risks Scale; measures individual variability in risk assessment; three scores are produced ("need for control", "self-confidence", "risk/thrill seeking"), all scores range from 0 to 100 with higher scores indicating a higher degree of the construct (e.g., higher risk/thrill seeking scores indicate a greater degree of risk/thrill seeking)

CONTACTS AND LOCATIONS:
Locations (1):
- US Army Aeromedical Research Laboratory, Fort Rucker, Alabama, United States

DOCUMENTS (1):
  • Informed Consent Form (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT03893032/ICF_000.pdf